CLINICAL TRIAL: NCT00015171
Title: CS1008 A&B Eff/Safety Trial of BUP/NX for the Treatment of Opiate Dependence
Brief Title: Buprenorphine and Naloxone for the Treatment of Opiate Dependence - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-5-0013-1; Y01-5-0013-1
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1999-01

CONDITIONS: Heroin Dependence; Substance-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Heroin Dependence; Substance-Related Disorders; Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is the use of buprenorphine/naloxone in treatment of opioid dependence.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and efficacy of a buprenorphine/naloxone combination tablet for opiate dependence treatment.

ELIGIBILITY:
Inclusion Criteria:

DSM-IV diagnosis of current opiate dependence males and non-pregnant, non-nursing female 18-59 yrs of age

Exclusion Criteria:

Any significant medical condition AST or ALT levels greater than 3x's the upper limit of normal level Current Axis I diagnosis other than opiate, caffeine or nicotine dependence

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-04; Primary Completion 1997-05 (Actual); Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
Craving
Drug use
Retention
Opioid withdrawal
Subjective rating

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States